CLINICAL TRIAL: NCT01963546
Title: Effects of Different Types of Anesthesia on Stress Response in Laparoscopic Gastric Bypass for Type 2 Diabetes Mellitus and the Effect of Dexmedetomidine on the Stress Response in Patients With Diabetic Undergoing Gastric-bypass Surgery
Brief Title: Effects of Different Types of Anesthesia on Stress Response in Laparoscopic Gastric Bypass for Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Wenbin Qie, Effects of Different Types of Anesthesia on Stress Response in Laparoscopic Gastric Bypass for Type 2 Diabetes Mellitus, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WQie
Record Dates: First submitted 2013-09-30; First posted 2013-10-16 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes; Stress; Anesthesia
Keywords: diabetic; laparoscopic gastric bypass surgery; stress response; anesthesia; dexmedetomidine
MeSH Terms: conditions — Diabetes Mellitus; Fractures, Stress | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Intravenous anesthesia (Other): We use total intravenous anesthesia to assess the stress response.
  Interventions: Other: different types of anesthesia
- Intravenous and Inhalation anesthesia (Other): We use intravenous and inhalation anesthesia during the surgery.
  Interventions: Other: different types of anesthesia
- Inhalation anesthesia (Other): We use inhalation anesthesia during the surgery.
  Interventions: Other: different types of anesthesia
- Dexmedetomidine (Experimental): the effect of dexmedetomidine on the stress responses generated by patients with diabetic given gastric-bypass surgery : Group A group given the best anesthetic technique from preliminary work + dexmedetomidine Dexmedetomidine as a inducer was given intravenous infusion loading dose 1.0μg/kg for 10min, maintained intravenous infusion by 0.4μg/kg/h.
  Group B group given the best anesthesia method from preliminary work(not using dexmedetomidine).
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Other: different types of anesthesia
  Arms: Inhalation anesthesia; Intravenous and Inhalation anesthesia; Intravenous anesthesia
Drug: Dexmedetomidine — After selecting the appropriate anesthesia method, assess the effect of dexmedetomidine on controlling stress response from diabetics undergoing laparoscopic gastric-bypass surgical.The stress indicators are the same as described above.
  Arms: Dexmedetomidine

SUMMARY:
General anesthesia can be considered as a combination of hypnosis, antinociception and immobility. Explore the effect of three kinds of anesthesia,that is the total intravenous anesthesia, inhalation anesthesia and inhalation and intravenous anesthesia on stress reactions generated by patients with diabetes conducted gastric - bypass surgery , and choose a best way from three kinds of anesthesia to control stress reaction of diabetics. After selecting the appropriate anesthesia method, assess the effect of dexmedetomidine on controlling stress response from diabetics undergoing laparoscopic gastric-bypass surgical.

DETAILED DESCRIPTION:
Research content and indicators

1. Preparation of serum: 3ml of blood were taken before induction of anesthesia (after entering the operating room), surgery began 1h, surgery began 2h, 24h after surgery, and placed at dry tube, centrifuged for 10min at 3000g after placing at room temperature for 2h , the resulting supernatant was subpassaged in tube, stored at -20℃ until analysis.
2. Indicators to detect in serum contained Tumor Necrosis Factor-α, Interleukin-6, Interleukin-10, plasma glucose, cortisol,insulin and c-peptide.
3. Record the vital signs.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists（ASA）Ⅰ ~ Ⅱpatients
* Type 2 Diabetes Mellitus patient undergoing Laparoscopic Gastric Bypass surgery
* between 18 and 60 years of age

Exclusion Criteria:

* A history of cardiopulmonary disease, liver and kidney dysfunction, abnormal coagulation
* Thyroid disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Stress Indicators | 72 hours
  We use different anesthesia method to assess the stress indicators,aiming to choose an apposite anesthesia to reduce stress response in laparoscopic gastric bypass for type 2 diabetes mellitus.The stress indicators include Tumor Necrosis Factor-α,Interleukin-10,Interleukin-6,C-peptide,Cortisol,Insulin and Adrenocorticotropic hormone.

SECONDARY OUTCOMES:
Vital Signs | during surgery
  We record blood pressure, heart rate, end-tidal carbon dioxide,mean arterial pressure at the time of intubation and 45min,90min when the surgery start.

CONTACTS AND LOCATIONS:
Overall Officials: Tu wei feng, Postdoctoral, Principal Investigator — The General Hospital Of Guangzhou Military Command
Locations (1):
- The General Hospital Of Guangzhou Military Command, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Cheng YC, Cheng XB, Li XJ, Wang FZ, Li ZK. Combined general and regional anesthesia and effects on immune function in patients with benign ovarian tumors treated by laparoscopic therapy. Int J Clin Exp Med. 2013 Sep 1;6(8):716-9. eCollection 2013. PMID 24040483
- [Background] Dell'Aquila AM, Ellger B. Perioperative glycemic control: what is worth the effort? Curr Opin Anaesthesiol. 2013 Aug;26(4):438-43. doi: 10.1097/ACO.0b013e328362d16a. PMID 23743557
- [Background] Ezhevskaya AA, Mlyavykh SG, Anderson DG. Effects of continuous epidural anesthesia and postoperative epidural analgesia on pain management and stress response in patients undergoing major spinal surgery. Spine (Phila Pa 1976). 2013 Jul 1;38(15):1324-30. doi: 10.1097/BRS.0b013e318290ff26. PMID 23514874
- [Background] Hadimioglu N, Ulugol H, Akbas H, Coskunfirat N, Ertug Z, Dinckan A. Combination of epidural anesthesia and general anesthesia attenuates stress response to renal transplantation surgery. Transplant Proc. 2012 Dec;44(10):2949-54. doi: 10.1016/j.transproceed.2012.08.004. PMID 23195004